CLINICAL TRIAL: NCT05155579
Title: A Phase Ib Trial to Evaluate the Safety and Immunogenicity of R21/Matrix-M in a Single and Two Vial Presentation, With Different Immunisation Schedules, and When Co-Administered With EPI Vaccines in African Children
Brief Title: Assessment of Safety and Immunogenicity of a Single Vial Presentation of R21/Matrix-M and Co-Administration With EPI Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Malaria Research and Training Center, Bamako, Mali (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VAC088
Record Dates: First submitted 2021-12-09; First posted 2021-12-13 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — Tetanus Toxoid; Hepatitis B Vaccines

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant, Investigator
Masking Description: For groups 1, 2 and 3, participants and investigators will be blinded to group allocation. Study staff involved in storage and preparation of the vaccine will be aware of vaccine assignment but these staff will play no other role in the study. The Sponsor team will remain blinded with the exception of designated members of the laboratory team that will perform the final evaluation of the data. For groups 4 and 5, no study staff or participants will be blinded as the number of vaccinations in each group is different. For group 6, no study staff or participants will be blinded as the schedule of vaccinations in each group is different.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- Groups 1a, 2a and 3a (Experimental): 60 children, aged 5-36 months, who will receive 4 doses of 5µg R21/50µg Matrix-M as a two vial formulation. The first three doses will be given one month apart, followed by a booster vaccination 12 months after the third dose. The age range of 5-36 months has been split into three groups to ensure an even age spread across age groups. Group 1a is 20 children aged 5-11 months, group 2a is 20 children aged 12-23 months, and group 3a is 20 children aged 24-36 months.
  Interventions: Biological: R21/Matrix-M - two vial formulation
- Group 1b, 2b and 3b (Experimental): 60 children, aged 5-36 months, who will receive 4 doses of 5µg R21/50µg Matrix-M as a single vial formulation. The first three doses will be given one month apart, followed by a booster vaccination 12 months after the third dose. The age range of 5-36 months has been split into three groups to ensure an even age spread across age groups. Group 1b is 20 children aged 5-11 months, group 2b is 20 children aged 12-23 months, and group 3b is 20 children aged 24-36 months.
  Interventions: Biological: R21/Matrix-M - single vial formulation
- Group 4a (Experimental): 150 participants, aged 6-7 months at the time of randomisation (to ensure third vaccination is given at approximately 9 months), who will receive 3 doses of 5µg R21/50µg Matrix-M one month apart. At the time of the third dose they will receive their measles-rubella and yellow fever vaccinations at the same time as R21/Matrix-M.
  Interventions: Biological: R21/Matrix-M - single vial formulation; Biological: Licensed vaccine - Measles-rubella; Biological: Licensed vaccine - Yellow fever
- Group 4b (Active Comparator): 150 participants, aged 6-7 months at the time of randomisation, who will receive a measles-rubella and yellow fever vaccination 2 months after randomisation.
  Interventions: Biological: Licensed vaccine - Measles-rubella; Biological: Licensed vaccine - Yellow fever
- Group 4c (Experimental): Group 4c is 50 participants, aged 6-7 months at the time of randomisation, who will receive 3 doses of 5µg R21/50µg Matrix-M one month apart.
  Interventions: Biological: R21/Matrix-M - single vial formulation
- Group 5a (Experimental): 30 children who will receive 3 doses of 5µg R21/50µg Matrix-M, pentavalent, rotavirus, pneumococcal and OPV vaccines at 6, 10 and 14 weeks of age. They will receive IPV two weeks following the third dose.
  Interventions: Biological: R21/Matrix-M - single vial formulation; Biological: Licensed vaccine - Pentavalent (diphtheria, tetanus, pertussis, hepatitis B and Hib); Biological: Licensed vaccine - Oral Polio Vaccine (OPV); Biological: Licensed vaccine - Rotavirus; Biological: Licensed vaccine - Pneumococcal vaccine; Biological: Licensed vaccine - Inactivated Polio Vaccine (IPV)
- Group 5b (Active Comparator): 30 children who will receive 3 doses of pentavalent, rotavirus, pneumococcal and OPV vaccines at 6, 10 and 14 weeks of age. They will receive IPV two weeks following the third dose.
  Interventions: Biological: Licensed vaccine - Pentavalent (diphtheria, tetanus, pertussis, hepatitis B and Hib); Biological: Licensed vaccine - Oral Polio Vaccine (OPV); Biological: Licensed vaccine - Rotavirus; Biological: Licensed vaccine - Pneumococcal vaccine; Biological: Licensed vaccine - Inactivated Polio Vaccine (IPV)
- Group 6a (Experimental): 30 children, aged 5-36 months, who will receive 3 doses of 5µg R21/50µg Matrix-M. The first two doses one month apart and the third dose 6 months after the first dose.
  Interventions: Biological: R21/Matrix-M - single vial formulation
- Group 6b (Experimental): 30 children, aged 5-36 months, who will receive 3 doses of 5µg R21/50µg Matrix-M. The first two doses one month apart and the third dose 12 months after the first dose.
  Interventions: Biological: R21/Matrix-M - single vial formulation

INTERVENTIONS:
Biological: R21/Matrix-M - single vial formulation — Adjuvanted malaria vaccine in a single vial formulation
  Arms: Group 1b, 2b and 3b; Group 4a; Group 4c; Group 5a; Group 6a; Group 6b
Biological: R21/Matrix-M - two vial formulation — Adjuvanted malaria vaccine in a double vial formulation
  Arms: Groups 1a, 2a and 3a
Biological: Licensed vaccine - Measles-rubella — Licensed vaccine part of the EPI vaccination schedule
  Arms: Group 4a; Group 4b
Biological: Licensed vaccine - Yellow fever — Licensed vaccine part of the EPI vaccination schedule
  Arms: Group 4a; Group 4b
Biological: Licensed vaccine - Pentavalent (diphtheria, tetanus, pertussis, hepatitis B and Hib) — Licensed vaccine part of the EPI vaccination schedule
  Arms: Group 5a; Group 5b
Biological: Licensed vaccine - Oral Polio Vaccine (OPV) — Licensed vaccine part of the EPI vaccination schedule
  Arms: Group 5a; Group 5b
Biological: Licensed vaccine - Rotavirus — Licensed vaccine part of the EPI vaccination schedule
  Arms: Group 5a; Group 5b
Biological: Licensed vaccine - Pneumococcal vaccine — Licensed vaccine part of the EPI vaccination schedule
  Arms: Group 5a; Group 5b
Biological: Licensed vaccine - Inactivated Polio Vaccine (IPV) — Licensed vaccine part of the EPI vaccination schedule
  Arms: Group 5a; Group 5b

SUMMARY:
This is a Phase Ib trial conducted in Bougouni, Mali to evaluate the safety and immunogenicity of R21/Matrix-M in a single and two vial presentation, with different immunisation schedules, and when co-administered with EPI vaccines in African children.

DETAILED DESCRIPTION:
This trial has six groups. This will be a double-blind, individually randomised trial, with 1:1 randomisation with the single or two vial presentation of R21/Matrix-M malaria vaccine for study groups 1, 2 and 3. Groups 1, 2 and 3 are to assess the safety and immunogenicity of R21/Matrix-M as a single vial formulation compared with a two-vial formulation, in children aged 5- 36 months, in a malaria endemic area. The age range of 5-36 months has been split into three groups to ensure an even age spread across age groups.

For groups 4 and 5, this is a randomised, open-label study to assess the safety and immunogenicity of R21/Matrix-M when co-administrated with various EPI vaccines at the relevant ages, in a malaria endemic area.

Group 6 is a randomised, open-label study to assess safety and immunogenicity of a delayed, third dose of R21/Matrix-M in 5-36 month old children, in a malaria endemic area.

For groups 1, 2, 3, 5 and 6, participants will be randomised 1:1. For group 4, participants will be randomised 3:3:1.

Approximately 590 children will be recruited across these six study groups.

The primary study objectives are:

Safety

* To assess the safety and reactogenicity of R21/Matrix-M, as a single- vial formulation in 5-36-month old African children.
* To assess the safety and reactogenicity of co-administration of R21/Matrix-M with the EPI vaccines given at 9 months, measles-rubella and yellow fever vaccines, in African children.
* To assess the safety and reactogenicity of co-administration of R21/Matrix-M with the EPI vaccines given at 6, 10 and 14 weeks of age, pentavalent and oral polio vaccine (OPV), in African children.

Immunogenicity

* To assess the immunogenicity of R21/Matrix-M, as a single- vial formulation in 5-36-month-old African children, compared with the two-vial formulation.
* To assess the immunogenicity of EPI vaccines given at 9 months, measles-rubella and yellow fever vaccines, when given with and without R21/Matrix-M
* To assess the immunogenicity of EPI vaccines given at 6, 10 and 14 weeks of age, pentavalent and oral polio vaccines, given as part of EPI at 6, 10 and 14 weeks of age, when given with and without R21/Matrix-M.

The secondary study objectives are:

* To assess the safety and reactogenicity of R21/Matrix-M, as a single- vial formulation in African children compared with the two-vial formulation.
* To assess the safety and reactogenicity of a delayed third dose of R21/Matrix-M in 5-36-month-old African children.
* To assess the immunogenicity of a delayed third dose of R21/Matrix-M in 5-36-month-old African children.

This trial is funded by the Serum Institute of India.

ELIGIBILITY:
Inclusion Criteria at study entry:

* Age:

  * Group 1: The child is 5-11 months of age at the time of randomization (i.e. up to the day before of their first birthday).
  * Group 2: The child is 12-23 months of age at the time of randomization (i.e. up to the day before of their second birthday).
  * Group 3: The child is 24-36 months of age at the time of randomization (i.e. up to the day of their third birthday).
  * Group 4: The child is 6-7 months of age at the time of randomization.
  * Group 5: The child is 6 weeks of age at the time of randomization and have not received any dose of the pentavalent vaccine, pneumococcal vaccine, rotavirus vaccine, IPV and only the first dose of the OPV.
  * Group 6: The child is aged 5-36 months at the time of their first vaccination
* Signed informed consent/thumb-printed and witnessed informed consent obtained from the parent(s)/guardian(s) of the child to join the trial.
* The investigator believes that the parents/guardians can and will comply with the requirements of the protocol if the child is enrolled in the study.
* The child is a permanent resident of the study area and likely to remain a resident for the duration of the trial.

Exclusion Criteria at study entry:

* The child has previously received a malaria vaccine.
* The child is enrolled in another malaria intervention trial that could interfere with the results of this study.
* The child has a history of allergic disease or reactions likely to be exacerbated by any component of the study vaccines.
* The child has a history of allergic reactions, significant IgE-mediated events or anaphylaxis to previous immunisations.
* The child has major congenital defects.
* The child has anaemia associated with clinical signs of symptoms of decompensation, or a haemoglobin of ≤7.4 g/dL.
* The child has had a blood transfusion within one month of enrolment.
* The child has been administered immunoglobulins and/or any blood products within the three months preceding the planned administration of the vaccine candidate.
* The child has malnutrition requiring hospital admission.
* The child has an acute or chronic, clinically significant pulmonary, cardiovascular, gastrointestinal, endocrine, neurological, skin, hepatic or renal functional abnormality, as determined by medical history, physical examination or laboratory tests.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV or asplenia.
* The child has received an investigational drug or vaccine other than the study vaccines within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* The child is currently participating in another clinical trial if likely to affect data interpretation of this trial
* The child has any significant disease, disorder or situation which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Clinically significant laboratory abnormality as judged by the study clinician
* For group 5 only: the child has received any dose of the pentavalent vaccine, pneumococcal vaccine, rotavirus vaccine, IPV or has received more than one dose of the OPV.

Exclusion criteria during the study (to be checked prior to each vaccination):

• Any significant disease, disorder or situation which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Ages: 6 Weeks to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 593 (Actual)
Dates: Start 2022-05-14 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Safety | 2 years
  Solicited adverse events:
  * Occurrence of solicited local reactogenicity signs and symptoms for 7 days following the vaccination.
  * Occurrence of solicited systemic reactogenicity signs and symptoms for 7 days following the vaccination.
  Unsolicited adverse events
  * Occurrence of unsolicited adverse events for 28 days following the vaccination. Laboratory adverse events
  * Change from baseline for safety laboratory measures thought to be clinically significant.
  Serious adverse events
  • Occurrence of serious adverse events for the whole study duration.
Immunogenicity | 2 years
  * To assess the humoral immunogenicity of R21/Matrix-M as a single- vial formulation in 5-36-month-old African children, compared with the two-vial formulation, 0, 30, 180 and 365 days after the administration of the third dose of R21/Matrix-M; and 0, 30, 180 and 365 days after the administration of a booster dose.
  * To assess the humoral immunogenicity of EPI vaccines given at 9 months, measles-rubella and yellow fever vaccines, when given with and without R21/Matrix-M, 0, 30, 180 and 360 days after the administration of the third dose of R21/Matrix-M
  * To assess the humoral immunogenicity of EPI vaccines given at 6, 10 and 14 weeks of age, pentavalent and oral polio vaccines, given as part of EPI at 6, 10 and 14 weeks of age, when given with and without R21/Matrix-M, 0, 30, 180 and 360 days after the administration of the third dose of R21/Matrix-M or the EPI vaccines.

SECONDARY OUTCOMES:
Safety of a delayed third dose | 2 years
  Solicited adverse events:
  * Occurrence of solicited local reactogenicity signs and symptoms for 7 days following the vaccination.
  * Occurrence of solicited systemic reactogenicity signs and symptoms for 7 days following the vaccination.
  Unsolicited adverse events
  * Occurrence of unsolicited adverse events for 28 days following the vaccination. Laboratory adverse events
  * Change from baseline for safety laboratory measures thought to be clinically significant.
  Serious adverse events
  • Occurrence of serious adverse events for the whole study duration.
Immunogenicity of a delayed third dose | 2 years
  • To assess the humoral immunogenicity of a delayed third dose of R21/Matrix-M in 5-36-month-old African children, at 30 and 180 days after administration of the second dose, and 0, 30, 180 and 360 days after the administration of the third dose of R21/Matrix-M

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Hill, Principal Investigator — University of Oxford
Locations (2):
- Malaria Research & Training Center, Department of Epidemiology of Parasitic Diseases, Faculty of Medicine, Pharmacy and Dentistry, University of Sciences Techniques and Technologies of Bamako, Bamako, Mali
- CCVTM, University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided